CLINICAL TRIAL: NCT05822492
Title: Comparison of the Effects of Anterior Quadratus Lumborum Block and Erector Spina Plane Block on Postoperative Acute Pain in Percutaneous Nephrolithotomy Surgery
Brief Title: Anterior Quadratus Lumborum Block Versus Erector Spina Plane Block in Percutaneous Nephrolithotomy Surgery
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cengiz KAYA, Principal Investigator, Clinical Professor, Ondokuz Mayıs University
Other Study IDs: PNLESPQLB2022
Record Dates: First submitted 2023-04-10; First posted 2023-04-20 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia; Analgesia; Patient Controlled Analgesia; Quadratus Lumborum Block; Erector Spina Plane Block
Keywords: Anesthesia; Analgesia; Percutaneous Nephrolithotomy Surgery; Patient controlled analgesia; Anterior quadratus lumborum block; Erector spina plane block
MeSH Terms: conditions — Agnosia | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group QLB3: Patients who applied the QLB3 block before PCNL surgery were included in this group.
  Interventions: Procedure: Group QLB3
- Group ESPB: Patients who applied ESP block before PCNL surgery were included in this group.
  Interventions: Procedure: Group ESPB
- Group Control: Patients who did not use any block before PCNL surgery were included in this group.
  Interventions: Other: Group Control

INTERVENTIONS:
Procedure: Group QLB3 — Patients who applied the QLB3 block before PCNL surgery were included in this group
  Multimodal analgesia protocol is applied to all patients undergoing PCNL surgery in our clinic. According to this protocol, patients are administered iv tenoxicam 20mg after induction of general anesthesia and iv paracetamol 1 gr intraoperatively. Postoperative analgesia: iv paracetamol 1gr every 8 hours and iv PCA of 0,2mg/ml morphine (the bolus dose is 20 mcg/kg, the lock-in time of 6-10 minutes, and the 4-hour limit is adjusted to be 80% of the calculated total dose). In cases where rescue analgesia is required (VAS score ≥4), 100 mg tramadol is administered to patients. The prophylaxis for postoperative nausea and vomiting (PONV) involved the routine administration of 8 mg IV dexamethasone to patients before induction and 0.15 mg/kg IV ondansetron 20 minutes before the end of the procedure.
  Other Names: Anterior Quadratus Lumborum Block (QLB3)
  Groups: Group QLB3
Procedure: Group ESPB — Patients who applied ESP block before PCNL surgery were included in this group
  Multimodal analgesia protocol is applied to all patients undergoing PCNL surgery in our clinic. According to this protocol, patients are administered iv tenoxicam 20mg after induction of general anesthesia and iv paracetamol 1 gr intraoperatively. Postoperative analgesia: iv paracetamol 1gr every 8 hours and iv PCA of 0,2mg/ml morphine (the bolus dose is 20 mcg/kg, the lock-in time of 6-10 minutes, and the 4-hour limit is adjusted to be 80% of the calculated total dose). In cases where rescue analgesia is required (VAS score ≥4), 100 mg tramadol is administered to patients. The prophylaxis for postoperative nausea and vomiting (PONV) involved the routine administration of 8 mg IV dexamethasone to patients before induction and 0.15 mg/kg IV ondansetron 20 minutes before the end of the procedure.
  Other Names: Erector spina plane block (ESPB)
  Groups: Group ESPB
Other: Group Control — Patients who did not use block before PCNL surgery were included in this group.
  Multimodal analgesia protocol is applied to all patients undergoing PCNL surgery in our clinic. According to this protocol, patients are administered iv tenoxicam 20mg after induction of general anesthesia and iv paracetamol 1 gr intraoperatively. Postoperative analgesia: iv paracetamol 1gr every 8 hours and iv PCA of 0,2mg/ml morphine (the bolus dose is 20 mcg/kg, the lock-in time of 6-10 minutes, and the 4-hour limit is adjusted to be 80% of the calculated total dose). In cases where rescue analgesia is required (VAS score ≥4), 100 mg tramadol is administered to patients. The prophylaxis for postoperative nausea and vomiting (PONV) involved the routine administration of 8 mg IV dexamethasone to patients before induction and 0.15 mg/kg IV ondansetron 20 minutes before the end of the procedure.
  Other Names: Control
  Groups: Group Control

SUMMARY:
In this study, it was aimed to evaluate the effects of anterior quadratus lumborum block (QLB3) and Erector Spina Plane Block (ESPB) on postoperative acute pain scores and opioid consumption in the first 24 hours in Percutaneous Nephrolithotomy Surgery

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is commonly used to treat large kidney stones. Patients usually complain of severe pain and discomfort postoperatively. Postoperative pain prolongs hospital stay, delays wound healing, increases infection rates, and increases the incidence of drug side effects.

Regional anesthesia is part of multimodal analgesia in treating postoperative pain. Facial plane blocks are among these procedures. Erector spina plane block (ESPB) is a peri-paravertebral regional anesthesia technique applied for the first time to treat thoracic neuropathic pain. In the literature, the effectiveness of upper abdomen and renal operations in pain management has been demonstrated. Quadratus lumborum block (QLB) was first described as an alternative to the transversus abdominis plane block. This block can be performed with three methods under ultrasound guidance. An anterior QLB (QLB3) block was used in this study. In this block, the local anesthetic drug is applied between the quadratus lumborum muscle and the psoas muscle fascia and spreads along the thoracolumbar fascia. This block provides anesthesia and analgesia in the T7-L1 dermatome area. QLB3 block has been applied in pyeloplasty, cholecystectomy, lower abdominal surgeries, cesarean sections, radical nephrectomy, and hip joint surgeries and provided adequate postoperative analgesia.

This study aimed to evaluate the effects of QLB3 block and ESPB block on pain scores and opioid consumption in patients undergoing PCNL.

Patients will be divided into three groups.

Group QLB3:

Patients who applied the OLB3 block and IV morphine-patient-controlled analgesia (PCA) before PCNL surgery were included in this group.

Group ESPB:

Patients who applied ESPB block and IV morphine-PCA before PCNL surgery were included in this group.

Group Control In this group, patients only applied general anesthesia and IV morphine-PCA.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* American Society of Anesthesiology score I-III patients scheduled for unilateral PCNL in elective conditions
* Patients with BMI <35 kg/m2

Exclusion Criteria:

* Pregnancy
* Conditions where regional anesthesia is contraindicated (coagulopathy, international normalized ratio abnormality, thrombocytopenia, infection at the injection site)
* History of hypersensitivity or allergy to local anesthetics
* Patients with psychiatric disorders
* Patients with musculoskeletal deformities
* Patients with alcohol-drug dependence
* Patients with cognitive dysfunction (patients incapable of evaluating the NRS score)
* Patients who did not give consent / did not want to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with undergoing percutaneous nephrolithotomy surgery,
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours after surgery | postoperative day 1
  Morphine consumption in the first 24 hours after surgery will be measured. Patients will be able to request opioids via a PCA device when their NRS score is ≥ 4.

SECONDARY OUTCOMES:
Postoperative pain scores | postoperative day 1
  Pain status at rest and while activity will be assessed by numeric rating scale (NRS) score at 0, 3, 6, 12, 18, and 24 hours after surgery. In addition, the time until the first analgesic requirement will be recorded. The NRS is an 11-point numeric scale that ranges from 0 to 10.
The postoperative nausea and vomiting (PONV) scores and the number of patients requiring antiemetic medication. | postoperative day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18, and 24 hours after extubation. If a score of 3 or more, ondansetron 4 mg IV will be administered and will repeat after 8 hours if required. The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once.
Intraoperative remifentanil consumption | The remifentanil consumption will be recorded from anesthesia induction until the patient is referred to the recovery unit, up to 150 minutes.
  The total amount of remifentanil consumed will be recorded.
The number of patient required rescue analgesia | postoperative day 1
  The number of patients requiring rescue analgesics will be recorded over 24 hours.
Time of first analgesic request | postoperative day 1
  Time at which the first analgesic is requested
The number of patients with complications | Postoperative 7 days on an average
  The number of patients has any complications -directly related to the block or the drug used in the block- will be recorded
The mean arterial pressure | The mean arterial pressure was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit, up to 180 minutes.
  The mean arterial pressure was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit.
The heart rate measurement | The heart rate was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit, up to 180 minutes.
  The heart rate was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit.

CONTACTS AND LOCATIONS:
Overall Officials: CENGIZ KAYA, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz mayıs Universty, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Dam M, Hansen CK, Poulsen TD, Azawi NH, Wolmarans M, Chan V, Laier GH, Bendtsen TF, Borglum J. Transmuscular quadratus lumborum block for percutaneous nephrolithotomy reduces opioid consumption and speeds ambulation and discharge from hospital: a single centre randomised controlled trial. Br J Anaesth. 2019 Aug;123(2):e350-e358. doi: 10.1016/j.bja.2019.04.054. Epub 2019 May 30. PMID 31153628
- [Background] Dam M, Moriggl B, Hansen CK, Hoermann R, Bendtsen TF, Borglum J. The Pathway of Injectate Spread With the Transmuscular Quadratus Lumborum Block: A Cadaver Study. Anesth Analg. 2017 Jul;125(1):303-312. doi: 10.1213/ANE.0000000000001922. PMID 28277325
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Elsharkawy H. Quadratus Lumborum Blocks. Adv Anesth. 2017;35(1):145-157. doi: 10.1016/j.aan.2017.07.007. Epub 2017 Oct 3. No abstract available. PMID 29103570
- [Background] Kilic E, Bulut E. Quadratus Lumborum Block III for Postoperative Pain After Percutaneous Nephrolithotomy. Turk J Anaesthesiol Reanim. 2018 Aug;46(4):272-275. doi: 10.5152/TJAR.2018.92331. Epub 2018 Aug 1. PMID 30140533
- [Derived] Turkan H, Kaya C, Turunc E, Dost B, Ustun YB. Effects of anterior quadratus lumborum block versus erector spinae plane block on postoperative acute pain in percutaneous nephrolithotomy: a prospective, observational study. BMC Anesthesiol. 2024 Sep 10;24(1):322. doi: 10.1186/s12871-024-02691-7. PMID 39256675